CLINICAL TRIAL: NCT00736008
Title: The Study Will Summarize the Clinical and Laboratory Data of All the Pediatric Patients Diagnosed With Thrombotic Events at the Pediatric Hematology Unit
Brief Title: Thrombophilic Risk Factors in Pediatric Patients Diagnosed at the Ha'Emek Medical Center
Status: Completed | Type: Observational
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Dr Koren Ariel, Head of Pediatric Hematology Unit and Pediatric Dpt B, HaEmek Medical Center, Israel
Other Study IDs: 0020-08-EMC
Record Dates: First submitted 2008-08-14; First posted 2008-08-15 (Estimated); Last update posted 2011-08-26 (Estimated); Status verified 2011-08

CONDITIONS: Thrombosis
Keywords: Factor V Leiden; Prothrombin Mutation; Hypercoagulability; Pediatrics
MeSH Terms: conditions — Thrombosis; Thrombophilia | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: Patients with thromboembolic events
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Data summary only

SUMMARY:
The study will assess the clinical and laboratory data of about 100 pediatric patients diagnosed and treated at the Pediatric Hematology Unit during the years 1980 until 2007 because of thrombotic events.

The results, the treatment given, and the outcome of the patients will be summarized.

ELIGIBILITY:
Inclusion Criteria:All the patients diagnosed since 1980.

Exclusion Criteria:Patients with insufficient data records.

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The population cohort will include about 100 patients diagnosed with thrombotic events at the Pediatric Hematology Unit
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2008-05; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carina Levin, MD, Principal Investigator — Pediatric Hematology Unit - Ha'Emek Medical Center - Afula - 18101 - Israel; Ayala Mari, Student, Principal Investigator — Pediatric Dpt B - Ha'Emek Medical Center - Afula - Israel
Locations (1):
- Pediatric Hematology Unit - Ha'Emek Medical Center, Afula, Afula, Israel